CLINICAL TRIAL: NCT04270240
Title: Can a New Scoring System Predict Hemodynamically Significant PDA Diagnosis and Treatment Requirement for Extremely Preterm Newborns Earlier
Brief Title: A NEW SCORING SYSTEM FOR PREDICTION OF PDA
Acronym: SIMPLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merih Cetinkaya, Neonatologist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: MAEEAH6725
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Patent Ductus Arteriosus; Prematurity; Extreme
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patent ductus arteriosus (PDA) is an important morbidity of that the diagnosis and treatment is controversy in premature infants. A number of scoring systems have been developed, including the findings of echocardiography on the diagnosis and treatment of PDA. This study aimed to develop a new clinical scoring system that will enable the rapid, standard and noninvasive evaluation of hemodynamically significant PDA earlier, without relying on echocardiographic findings in premature babies with extremely low birth weight, and to determine the role of this scoring system in early diagnosis and treatment.

DETAILED DESCRIPTION:
This study aimed to develop a new clinical scoring system that will enable the rapid, standard and noninvasive evaluation of hemodynamically significant PDA earlier, without relying on echocardiographic findings in premature babies with extremely low birth weight, and to determine the role of this scoring system in early diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* informed consent obtained from parents
* extremely preterm infants
* infants born before 28 gestational week

Exclusion Criteria:

* lack of informed consent
* chromosomal abnormality
* cardiovascular abnormality

Max Age: 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants who born before 28 gestational week and under 1000g of weight will be included.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Patent Ductus Arteriosus | 7 days
  number of participants who diagnosed for hemodynamically significant PDA and had an elevated score of the newly developed system by us.

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Yilmaz Semerci, Istanbul, Turkey (Türkiye)